CLINICAL TRIAL: NCT04350619
Title: Promote Personalized Medicine Based on Diagnostic Genomic Tools in Order to Innovate in the Early Detection of Child Deafness in the SUDOE Space (European International Project)
Brief Title: NGS Assessment of Congenitally Deafned Children and Neonatal Deafness Screnning
Acronym: GHELP
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Collaborators: Instituto de Salud Pública y Laboral de Navarra (Unknown); Biogipuzkoa Health Research Institute (Other); DREAMgenics S.L. (Unknown); Hospital CUF Porto, S.A. (Unknown); Centro Hospitalar de Lisboa Central (Other); University Hospital, Montpellier (Other); University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: GHELP
Record Dates: First submitted 2020-03-30; First posted 2020-04-17 (Actual); Last update posted 2020-04-17 (Actual); Status verified 2020-03

CONDITIONS: Congenital Deafness; Suspicion of Congenital Deafness
Keywords: Deafness; child
MeSH Terms: conditions — Deafness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood sample for genetic study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Genetic study in retrospective and prospective groups: Genetic screening using NGS technique in a retrospective and prospective groups. No therapeutic intervention
  Interventions: Other: Genetic screening. No therapeutic intervention

INTERVENTIONS:
Other: Genetic screening. No therapeutic intervention — Genetic screening using NGS technique. No therapeutic intervention

SUMMARY:
To assess the diagnostic value of NGS screnning in prelingually deafned children using a new designed chip, and to evaluate its interest in a the neonatal screening program for ddetecting congenitally deafned children.

DETAILED DESCRIPTION:
The aim of the study is to evaluate the diagnostic value of a new panel of gene in NGS study in children presenting :

1. A congenitally deafness : it is a retrospective study in children aged 0 to 17 yrs with hearing thresholds over 40 dB in the best ear using adapted audiometric assessment,
2. A suspicion of deafness in babies aged 0 to 6 months having an abnormal response after otoacoustic emissions and automated ABR assessment.

The main outcomes studied will be the finding of a pathogenic mutation (or several mutations).

ELIGIBILITY:
Inclusion Criteria:

* Retropective study

Inclusion criteria:

* Age of onset of deafness between 0 and 17 years
* With a hearing loss of one or two senses with, on the ear most affected, a hearing loss more than 40 dB in mean audiometric loss in behavioural audiometry
* Availability of detailed information in Appendix 1: History, history and course of disease, associated symptoms, otoscopy data, radiology, treatments and hearing aids implemented.
* Availability of DNA samples stored in an existing collection.
* Consent to participate in the study (non-opposition) by the legal representative

Exclusion Criteria:

* Exclusion criteria:

  * Child with a known cause of observed deafness (meningitis, post-surgery or drug iatrogenic, trauma, infections, tumor)
  * Family not willing to participate in the study

Prospective study

Inclusion criteria:

* Age of the child 0 to 6 months including corrected age having had on at least one of the two ears a lack of acoustic otoemissions and a lack of response in automated PEA, and a threshold of PEA at least on one ear at more than 40 dB.
* Availability of detailed information in Appendix 2: Personal history, family history of deafness, associated symptoms, tympanometry, otoscopy data, neonatal deafness test data.
* Collection of the consent of the legal representative

Exclusion criteria:

· Family not willing to participate in the study

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: There are 2 groups: retrospective and prospective which their characteristiques are described in the previous eligibility criteria.
Sampling Method: Probability Sample
Enrollment: 220 (Estimated)
Dates: Start 2020-04-30 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
Prevalence of mutation | 1 day
  It will realized the extraction blood sample in the same day and clinical information will be collected also.

SECONDARY OUTCOMES:
Phenotyping the mutation | 1 day
  Clinical information for each patient will be define for the following variables: age and gender, medical antecedents, audiometric data, other syndromic syntomps, ear radiologic data and type of treatment for treating the hearing loss.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Mondain, ENT, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Chu Montpellier, Montpellier, France